CLINICAL TRIAL: NCT02619175
Title: Characteristics of Balance Control to Unexpected Loss of Balance During Standing and Walking in Post-stroke Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nachum Soroker, MD (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor-Investigator, Nachum Soroker, MD, head, Department of neurologic rehabilitation, Loewenstein rehabilitation hospital, Raanana,Israel, Loewenstein Hospital
Organization: Loewenstein Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: loe150021ctil
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor

ARMS (2):
- Perturbation-based balance training (Experimental): perturbation-based balance training while standing and walking on the BalanceTutor (MediTouch).
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  Interventions: Device: Stroke Subjects Perturbation-Based Balance Training
- Weight shifting and gait training (Active Comparator): Balance and gait training without external perturbations. Voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill.
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  Interventions: Device: Stroke Subjects Weight Shifting and Gait training

INTERVENTIONS:
Device: Stroke Subjects Perturbation-Based Balance Training
  Arms: Perturbation-based balance training
Device: Stroke Subjects Weight Shifting and Gait training
  Arms: Weight shifting and gait training

SUMMARY:
aim: To examine the effect of a perturbation-based balance training on balance reaction characteristics in post stroke individuals.

DETAILED DESCRIPTION:
60 stroke subjects from the neurology rehabilitation unit at Loewenstein hospital will be randomly allocated to one of two groups: 1) perturbations based balance training 2) weight shifting and gait training without external perturbations (control).

Group 1 - Perturbations based balance training Subjects will complete a perturbation based balance training while standing and walking on the BalanceTutor (MediTouch). Perturbation level will be individually adjusted and progressed according to subject's abilities. Progression occurs by increasing perturbation level (increase distance, velocity and acceleration). At each practiced level subjects will be exposed to random right/left/forward/backward unannounced platform translations while standing and to right/left perturbations (in defined events in gait cycle) while walking. In order to examine adaptation to repeated perturbations, kinematic data will be collected in the first session.

Group 2 - Weight shifting and gait training Subjects will complete a balance training program that includes voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill. Weight shifting toward a target will be adjusted and progressed according to subject's abilities. Progression in difficulty level will occur by increasing the distance to target without changing the base of support. At each practiced level weight shifting will be conducted to right/left/forward/backward directions. In the gait part of the session, subjects will be asked to walk at their preferred treadmill walking speed.

Subjects in both groups will complete 10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes and will include practice in standing and walking. Subject's activities will be documented in each session in both groups. Furthermore, in each session subjects will be asked to rate their perceived level of challenge on a 0-10 scale.

Pre- and post-intervention measurements will be conducted. A follow-up measurement will be conducted 3-6 weeks post intervention.

The following measurements will be administered:

1)Compensatory balance reaction kinematic measurement:

Compensatory balance reactions will be measured using the BalanceTutor (MediTouch). The BalanceTutor is a mechatronic device consisting of a computerized treadmill with a horizontal movable platform and an operator station. Measurements will be taken in two conditions:

Standing. Subjects will be instructed to stand and will be exposed to random unexpected platform translations. The platform translations will be increased systematically and controlled. The increases in platform translation will be adjusted by the examiner to the subject's ability to recover from perturbations. Participants will be asked to respond in a "natural" manner to perturbations.

Walking. Subjects will be instructed to walk comfortably (self-paced) on the treadmill, and will be exposed to random unexpected platform translations. The platform translations will be increased systematically and controlled and will be adjusted by the examiner to the subject's ability to recover from perturbations. Compensatory balance reaction characteristics (reaction time, swing time, compensatory step time, step length etc.) will be collected through a three-dimensional motion analysis system. During examination subjects will wear a loose safety harness that will prevent a fall and yet allow the execution of balance recovery reactions.

In addition, clinical measures will be used: Berg Balance Scale, 6 minute walk test, 10 meter walk test, the Fugl-Meyer test for motor recovery after stroke and the ABC (Activities-specific Balance Confidence) scale. Normalized lesion data will be computed using the ABLE module within MEDx software (Medical Numerics).

ELIGIBILITY:
Inclusion Criteria:

For measurements taken while standing, post stroke subjects will meet the criteria of being able to stand independently or with supervision for at least 2 minutes.

For measurements taken while walking, post stroke subjects will meet the criteria of being able to walk for at least 10 meter with supervision/independently without walking aids.

* 3 weeks-6 months post stroke (hemorrhage/infarct)
* First stroke
* Age 25-75 years
* Able to understand research instructions
* Stable clinical/metabolic state

Exclusion Criteria:

* - A history of neurological diseases amongst peripheral neuropathy
* Significant skeletal system diseases, such as severe osteoporosis
* Uncontrolled atrial fibrillation
* Unstable ischemic heart disease
* Significant visual deficiency
* Dizziness
* Pregnancy
* Body weight above 135 kg

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: nachum Soroker, Principal Investigator — Loewenstein rehabilitation hospital, Raanana, ISRAEL
Locations (1):
- Loewenstein hospital, Raanana, Israel

REFERENCES:
- [Derived] Handelzalts S, Steinberg-Henn F, Farquhar J, Shkedy Rabani A, Levy S, Riemer R, Soroker N, Melzer I. Temporal But Not Spatial Gait Parameters Associated With Lower Balance Capacity in Moderate-High Functioning Persons With Stroke. J Neurol Phys Ther. 2021 Oct 1;45(4):301-309. doi: 10.1097/NPT.0000000000000368. PMID 34369447

RESULTS

PARTICIPANT FLOW:
Groups:
- Perturbation-based Balance Training, Stroke Subjects: perturbation-based balance training while standing and walking on the BalanceTutor (MediTouch).
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  BalanceTutor
- Weight Shifting and Gait Training, Stroke Subjects: Balance and gait training without external perturbations. Voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill.
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  posturograph
Period: Overall Study
Arm/Group | Perturbation-based Balance Training, Stroke Subjects | Weight Shifting and Gait Training, Stroke Subjects
Started | 18 | 16
Completed | 16 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — foot pain | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Perturbation-based Balance Training: perturbation-based balance training while standing and walking on the BalanceTutor (MediTouch).
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  BalanceTutor
- Weight Shifting and Gait Training: Balance and gait training without external perturbations. Voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill.
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  posturograph
- Total: Total of all reporting groups
Arm/Group | Perturbation-based Balance Training | Weight Shifting and Gait Training | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.7) | 60.4 (10.1) | 61.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Days post stroke [Mean (Standard Deviation); unit: days] | 40.6 (17.0) | 43.7 (19.7) | 42.0 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Compensatory Step Execution Time
Description: Will be calculated as the time from platform perturbation to foot contact using a 3D motion analysis system.
  Step execution time in response to surface translations toward the non-paretic side.
Time Frame: 1-5 days before the first session of intervention and 1-5 days after the last session of intervention.
Population: Analysis was conducted for step responses at perturbation level 3, since step responses were not frequently induced at low perturbation intensities and most subjects were not able to recover balance loss at higher perturbation intensities. Data represent subjects who reached intensity 3 without a fall in previous intensities (n=13 and n=8).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Perturbation-based Balance Training | Weight Shifting and Gait Training
Number analyzed (Participants) | 13 | 8
msec | -119.7 (236.6) | -4.2 (44.4)

2. Primary Outcome: Change in Compensatory Step Velocity
Description: will be calculated from step length and step swing time data, using a 3D motion analysis system.
  Step velocity in response to surface translations toward the non-paretic side.
Time Frame: 1-3 days before the first session of intervention and 1-3 days after the last session of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Perturbation Based Balance Training: perturbation-based balance training while standing and walking on the BalanceTutor (MediTouch).
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  BalanceTutor
- Weight-shifting and Gait Training: Balance and gait training without external perturbations. Voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill.
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  posturograph
Arm/Group | Perturbation Based Balance Training | Weight-shifting and Gait Training
Number analyzed (Participants) | 13 | 8
m/sec | 0.05 (0.2) | -0.05 (0.08)

3. Secondary Outcome: Change in Berg Balance Scale Score
Description: A 14-item objective measure (ordinal scale) designed to assess static balance and fall risk.
  Minimus score =0, Maximal score=56. Higher values represent a better outcome.
Time Frame: 1-3 days before the first session of intervention and 1-3 days after the last session of intervention.
Measure: Mean (Standard Deviation); unit: units on a scale 0-56.
Arm/Group | Perturbation-based Balance Training, Stroke Subjects | Weight Shifting and Gait Training, Stroke Subjects
Number analyzed (Participants) | 16 | 16
units on a scale 0-56. | 5.7 (3.9) | 5.8 (5.6)

4. Secondary Outcome: Change in Fall Threshold
Description: The perturbation level at which the subject lost balance and fell into the safety harness. Score on a scale (1-7). Each unit represents the perturbation intensity where the subject was unable to recover balance and fell into harness system. Higher values represent a better outcome.
Time Frame: 1-3 days before the first session of intervention and 1-3 days after the last session of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perturbation Based Balance Training | Weight Shifting and Gait Training
Number analyzed (Participants) | 16 | 16
score on a scale | 1.93 (1.6) | 1.12 (1.8)

5. Secondary Outcome: Change in Activities-specific Balance Confidence (ABC) Scale
Description: A self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. Score on a scale (0-100). Higher values represent a better outcome.
Time Frame: 1-3 days before the first session of intervention and 1-3 days after the last session of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perturbation-based Balance Training | Weight Shifting and Gait Training
Number analyzed (Participants) | 16 | 16
score on a scale | 17.9 (16.01) | 4.1 (9.23)

ADVERSE EVENTS:
Time Frame: from pre-intervention assessment until post-intervention assessment (1 month)
Groups:
- BalanceTutor: perturbation-based balance training while standing and walking on the BalanceTutor (MediTouch).
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  BalanceTutor
- Posturograph: Balance and gait training without external perturbations. Voluntary weight shifting while standing on a computerized posturography (NeuroCom) and walking on a treadmill.
  10-12 training sessions, 4-5 per week for 3 weeks. Each session will last 30 minutes.
  posturograph
Arm/Group | BalanceTutor | Posturograph
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 1/18 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BalanceTutor (N=18) | Posturograph (N=16)
foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT02619175/Prot_SAP_000.pdf